CLINICAL TRIAL: NCT03474965
Title: A Phase 2,Multicenter,Open-Label Study to Assess Appropriate Dosing and to Evaluate Safety of Crizanlizumab,With or Without Hydroxyurea/Hydroxycarbamide,in Sequential,Descending Age Groups of Pediatric Sickle Cell Disease Patients With Vaso-Occlusive Crisis
Brief Title: Study of Dose Confirmation and Safety of Crizanlizumab in Pediatric Sickle Cell Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSEG101B2201; 2017-001747-12 (EudraCT Number)
Record Dates: First submitted 2018-03-16; First posted 2018-03-23 (Actual); Results first posted 2025-07-20 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Sickle Cell Disease (SCD)
Keywords: SEG101; Sickle cell disease; SCD; crizanlizumab; pediatric; pharmacokinetic; P-selectin; Covid-19; Coronavirus disease 2019
MeSH Terms: conditions — Anemia, Sickle Cell; COVID-19 | interventions — crizanlizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Crizanlizumab (Experimental): SEG101 (crizanlizumab) 5 mg/kg or 8 mg/kg i.v. administered on Week 1 Day 1, Week3 Day 1 and Day 1 of every 4-week cycle for up to 2 years. The initial dose of crizanlizumab was 5 mg/kg dose for Group 1 and Group 2 Part A. It was later adjusted to 8.5 mg/kg for Group 2 and 3 based on final dose confirmation from emerging PK data analysis and safety considerations determined in Part A of the study.
  Interventions: Drug: Crizanlizumab

INTERVENTIONS:
Drug: Crizanlizumab — Crizanlizumab (SEG101) is a concentrate for solution for infusion, i.v. use. Supplied in single use 10 mL vials at a concentration of 10 mg/mL. One vial contains 100 mg of crizanlizumab.
  Other Names: SEG101

SUMMARY:
The purpose of this study was to confirm and to establish appropriate dosing and to evaluate the safety in pediatric participants ages 2 to <18 years with a history of Vaso-Occlusive Crisis (VOC) with or without Hydroxyurea/Hydroxycarbamide (HU/HC), receiving crizanlizumab for 2 years. The efficacy and safety of crizanlizumab was previously demonstrated in adults with sickle cell disease. The approach was to extrapolate from the pharmacokinetics (PK)/pharmacodynamics (PD) already established in the adult population. The study was designed as a Phase II, multicenter, open-label study.

DETAILED DESCRIPTION:
This was an open-label, single-arm study of crizanlizumab in sickle-cell disease (SCD) pediatric participants.

This study consisted of 2 parts, Part A and Part B. In Part A, the dose for 3 age groups (see groups below), was first confirmed on the basis of single and multiple dose (steady state) PK data and key safety data from an initial subgroup of participants. In Part B, safety and efficacy were collected from additional participants from 6 to <18 years (Groups 1 and 2, only).

At least 100 participants were planned to be enrolled in the trial in total, split in 3 age groups:

* Group 1 (age 12 to <18 years): at least 26 participants (≥8 in Part A and ≥18 in Part B),
* Group 2 (age 6 to <12 years): at least 26 participants (≥8 in Part A and ≥18 in Part B),
* Group 3 (age 2 to <6 years): at least 8 participants (≥8 Part A). Crizanlizumab was administered every 4 weeks with a loading dose 2 weeks after the first dosing (i.e., by i.v. infusion) on Week 1 Day 1, Week 3 Day 1, and then day 1 of every fourth week) for up to 2 years. The initial dose of crizanlizumab was 5 mg/kg dose for Group 1 and Group 2 Part A. It was later adjusted to 8.5 mg/kg for Group 2 and 3 based on final dose confirmation from emerging PK data analysis and safety considerations determined in Part A of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ages 2 to <18 years
2. Confirmed diagnosis of SCD (any genotype including HbSS, HbSC, HbSβ0-thalassemia, HbSβ+-thalassemia patients, and others) by hemoglobin electrophoresis or/and high-performance liquid chromatography (HPLC) [performed locally]. Confirmation of diagnosis by two accepted methods is recommended.
3. Experienced at least 1 VOC within the preceding 12 months prior to screening, as determined by medical history. Prior VOC must have resolved at least 7 days prior to the first dose in the study and must include all the following: a.the occurrence of appropriate symptoms (see VOC definition in Section 7.2.1.1), b.either a visit to a medical facility or healthcare professional, c.receipt of oral/parenteral opioid or parenteral NSAIDs
4. If receiving HU/HC, L-glutamine or erythropoietin stimulating agent, must have been receiving the drug consistently for at least 6 months prior to screening and plan to continue taking it at the same dose and schedule during the trial. Patients who have not been receiving such drugs must have been off them for at least 6 months prior to screening. . Dose alterations of HU/HC, L-glutamine or erythropoietin stimulating agent during Part A are not allowed, and if this occurs, the participant will enter directly to Part B.
5. Received standard age-appropriate care for SCD, including penicillin prophylaxis, pneumococcal immunization, and parental education.
6. Performance status: Karnofsky ≥ 50% for patients >10 years of age, and Lansky ≥ 50 for patients ≤ 10 years of age.
7. Patient must meet the following laboratory values prior to Week 1 Day 1: Absolute Neutrophil Count ≥1.0 x 109/L , Platelets ≥75 x 109/L, Hemoglobin (Hgb) > 5.5 g/dL
8. Patient must have adequate renal and hepatic function as defined:Estimated Glomerular filtration rate (eGFR) ≥ 75 mL/min/1.73 m2 using Schwartz formula, Direct (conjugated) bilirubin ≤ 2.0 x ULN, Alanine transaminase (ALT) ≤ 3.0 x ULN,
9. Transcranial Doppler (TCD) for patients aged 2 to < 16 years at time of screening, with HbSS, HbSβ0-thalassemia, and HbSD disease indicating low risk for stroke (per investigator). Please refer to Section 7.2.2.6 for details
10. Written informed consent/assent, according to local guidelines, signed by the patient and / or by the parents or legal guardian prior to any study related screening procedures are performed.
11. Female of non-childbearing potential or with negative serum pregnancy test on Screening and a negative urine pregnancy test (dipstick) prior to dosing on Day 1.

Exclusion Criteria:

1. History of stem cell transplant.
2. Received any blood products within 30 days prior to Week 1 Day 1 dosing.
3. Plan to participate in a chronic transfusion program (pre-planned series of transfusions for prophylactic purposes) or undergo exchange transfusions/plasmapheresis during the study. Patients requiring episodic transfusion (simple or exchange) in response to worsened anemia or VOC are permitted.
4. Patients with bleeding disorders

6.Contraindication or hypersensitivity to any drug from similar class as study drug or to any excipients of the study drug formulation.

7.History of severe hypersensitivity reaction to other monoclonal antibodies, which in the opinion of the investigator may pose an increased risk of serious infusion reaction 8.Received a monoclonal antibody or immunoglobulin-based therapy within 6 months of Screening, or has documented immunogenicity to a prior monoclonal antibody.

9.Received active treatment on another investigational trial within 30 days (or 5 half -lives of that agent, whichever is greater) prior to Screening or plans to participate in another investigational drug trial.

10.Pregnant females or females who have given birth within the past 90 days or who are breastfeeding.

11. Any documented history of a clinical stroke or intracranial hemorrhage, or an uninvestigated neurologic finding within the past 12 months. Silent infarcts (only present on imaging) are not excluding patients from study participation 12.Any abnormal TCD within the past 12 months. 13.Use of therapeutic anticoagulation (prophylactic doses permitted) or antiplatelet therapy (other than aspirin) within the 10 days prior to Week 1 Day 1 dosing.

14.Hospitalized within 7 days prior to Week 1 Day 1 dosing. 15.Planning to undergo a major surgical procedure during the duration of the study.

16.Planning to initiate or terminate HU/HC or L-glutamine while on study (except if needed to terminate for safety reasons).

17.Patient with active human immunodeficiency virus (HIV) infection (detectable viral load).

18.Patients with known active Hepatitis B infection. 19.Patients with known Hepatitis C history. 20.Significant active infection or immune deficiency (including chronic use of immunosuppressive drugs) in the opinion of the investigator.

21.Malignant disease. Exceptions to this exclusion include the following: malignancies that were treated curatively and have not recurred within 2 years prior to study treatment; any completely resected carcinoma in situ.

22.Has a serious mental or physical illness, which, in the opinion of the Investigator would compromise participation in the study.

23.Any condition which, in the opinion of the investigator, is likely to interfere with the successful collection of the measurements required for the study 24.Resting QTcF ≥450 msec at pretreatment (baseline) for patients under 12 years of age and ≥450 msec for males and ≥460 msec for female patients 12 years and older.

25.Cardiac or cardiac repolarization abnormality, including any of the following: a. History of myocardial infarction (MI), uncontrolled congestive heart failure, unstable angina, or coronary bypass graft (CABG) within 6 months prior to starting study treatment, b. Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high-grade AV block (bifascicular block, Mobitz Type II, and third degree AV block), c. Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome ( Risk factors for Torsade de Pointes (TdP), including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/ symptomatic bradycardia, Inability to determine the QTcF).

26. Sexually active females who are unwilling to comply with reliable method of birth control until 15 weeks following last dose of study drug.

28.Not able to understand and to comply with study instructions and requirements.

29.Patients who are an employee of the sponsor or investigator or otherwise dependent on them.

30.Patients who are committed to an institution by virtue of an order issued either by the judicial or the administrative authorities.

31.Patients who received prior crizanlizumab treatment and/or other selectin targeting agents are not allowed 32.Patients having taken voxelotor less than 30 days prior to Screening, or planning to take voxelotor while on study are not allowed.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 117 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (35):
- United States (12):
  - University Of Alabama, Birmingham, Alabama
  - Childrens National Hospital, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Joe DiMaggio Childrens Hospital, Hollywood, Florida
  - Childrens Healthcare of Atlanta, Atlanta, Georgia
  - Childrens Hosp Boston Dept of Hematology, Boston, Massachusetts
  - Childrens Hospital at Montefiore, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Childrens Hospital Of Philadelphia, Philadelphia, Pennsylvania
  - Medical Uni of South Carolina, Charleston, South Carolina
  - Cook Childrens Medical Center, Fort Worth, Texas
- Belgium (3):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Laken
  - Novartis Investigative Site, Liège
- Brazil (3):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Ribeirão Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Novartis Investigative Site, Montreal, Quebec, Canada
- Colombia (2):
  - Novartis Investigative Site, Cali, Valle del Cauca Department
  - Novartis Investigative Site, Montería
- Novartis Investigative Site, Paris, France
- Novartis Investigative Site, Heidelberg, Germany
- Novartis Investigative Site, Nagpur, Maharashtra, India
- Italy (2):
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Orbassano, TO
- Lebanon (2):
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, Tripoli
- Novartis Investigative Site, Muscat, Oman
- Spain (3):
  - Novartis Investigative Site, Palma de Mallorca, Balearic Islands
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Mersin
- Novartis Investigative Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- [Derived] Del Pozo Martin Y. 2021 ASH annual meeting. Lancet Haematol. 2022 Feb;9(2):e92-e93. doi: 10.1016/S2352-3026(21)00384-7. Epub 2021 Dec 16. No abstract available. PMID 34922648
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2606

RESULTS

PARTICIPANT FLOW:
Groups:
- Age 12 to <18 Years, 5 mg/kg: Age 12 to <18 years, 5 mg/kg
- Age 6 to <12 Years, 5 mg/kg: Age 6 to <12 years, 5 mg/kg
- Age 6 to <12 Years, 8.5 mg/kg: Age 6 to <12 years, 8.5 mg/kg
- Age 2 to <6 Years, 8.5 mg/kg: Age 2 to <6 years, 8.5 mg/kg
Period: Overall Study
Arm/Group | Age 12 to <18 Years, 5 mg/kg | Age 6 to <12 Years, 5 mg/kg | Age 6 to <12 Years, 8.5 mg/kg | Age 2 to <6 Years, 8.5 mg/kg
Started | 50 | 13 | 40 | 14
Completed | 33 | 10 | 29 | 11
Not Completed | 17 | 3 | 11 | 3
Not completed — Pregnancy | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 1
Not completed — Physician Decision | 3 | 1 | 2 | 0
Not completed — Participant Decision | 7 | 0 | 1 | 0
Not completed — Guardian Decision | 4 | 2 | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Age 12 to <18 Years, 5 mg/kg | Age 6 to <12 Years, 5 mg/kg | Age 6 to <12 Years, 8.5 mg/kg | Age 2 to <6 Years, 8.5 mg/kg | Total
Number analyzed (Participants) | 50 | 13 | 40 | 14 | 117
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50 | 13 | 40 | 14 | 117
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 15.00 (1.921) | 8.87 (1.745) | 9.29 (1.614) | 4.81 (0.868) | 11.15 (3.983)
Age, Customized [Count of Participants; unit: Participants]
  0 - <28 d | 0 | 0 | 0 | 0 | 0
  28 d - <2 y | 0 | 0 | 0 | 0 | 0
  2 y - <12 y | 0 | 13 | 40 | 14 | 67
  12 y - <18 y | 50 | 0 | 0 | 0 | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 5 | 17 | 5 | 56
  Male | 21 | 8 | 23 | 9 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 3 | 4 | 7
  Asian | 7 | 0 | 3 | 0 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 32 | 7 | 19 | 8 | 66
  White | 11 | 4 | 13 | 2 | 30
  More than one race | 0 | 2 | 2 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): AUCd15 of Crizanlizumab After First Dose - Part A
Description: The area under the curve (AUC) from time zero to the last measurable concentration sampling time (tlast) (mass x time x volume-1) following the first dose. AUCd15 was calculated based on serum concentrations of crizanlizumab.
Time Frame: Day 1 to Day 15
Population: Pharmacokinetic analysis set 1 - for treated participants with a valid measurement without a protocol deviation with impact.
Measure: Mean (Standard Deviation); unit: hr*ug/mL
Arm/Group | Age 12 to <18 Years, 5 mg/kg | Age 6 to <12 Years, 5 mg/kg | Age 6 to <12 Years, 8.5 mg/kg | Age 2 to <6 Years, 8.5 mg/kg
Number analyzed (Participants) | 10 | 11 | 13 | 10
hr*ug/mL | 10500 (2290) | 8180 (1620) | 20600 (4530) | 14400 (3990)

2. Primary Outcome: Pharmacokinetics (PK) - AUCtau for Serum Crizanlizumab After Multiple Doses - Part A - Steady State
Description: The AUC calculated to the end of a dosing interval (tau) at steady-state (amount x time x volume-1).
Time Frame: Week 15 - Steady state
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr*ug/mL
Arm/Group | Age 12 to <18 Years, 5 mg/kg | Age 6 to <12 Years, 5 mg/kg | Age 6 to <12 Years, 8.5 mg/kg | Age 2 to <6 Years, 8.5 mg/kg
Number analyzed (Participants) | 7 | 6 | 11 | 12
hr*ug/mL | 15800 (2080) | 14800 (3770) | 35700 (8100) | 22100 (6200)

3. Primary Outcome: Pharmacokinetics (PK) - Cmax for Crizanlizumab After First Dose and Multiple Doses - Part A - Steady State
Description: The maximum (peak) observed, serum, drug concentration after single or multiple dose administration (mass x volume-1)
Time Frame: Week 1 (after first dose) and Week 15 (steady state)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Age 12 to <18 Years, 5 mg/kg | Age 6 to <12 Years, 5 mg/kg | Age 6 to <12 Years, 8.5 mg/kg | Age 2 to <6 Years, 8.5 mg/kg
Number analyzed (Participants) | 11 | 11 | 13 | 12
ug/mL
  PK Single Dose (Week 1) (n=11,11,13,10): number analyzed (Participants) | 11 | 11 | 13 | 10
  PK Single Dose (Week 1) (n=11,11,13,10) | 80.5 (17.7) | 65.9 (11.3) | 175 (36.0) | 110 (37.3)
  PK Multiple Dose - Week 15 (Steady state) (n=7,8,12,12): number analyzed (Participants) | 7 | 8 | 12 | 12
  PK Multiple Dose - Week 15 (Steady state) (n=7,8,12,12) | 95.6 (26.6) | 77.5 (19.0) | 171 (35.3) | 111 (27.4)

4. Primary Outcome: Pharmacodynamics (PD) - P-selectin Inhibition Parameters for Crizanlizumab After First Dose - Part A - AUCd15
Description: The AUC from time zero to the last measurable concentration sampling time (tlast) (mass x time x volume-1) following the first dose. AUCd15 was calculated based on P-selectin inhibition curves.
Time Frame: Day 1 to Day 15
Population: Pharmacodynamic analysis set 1 - for treated participants with a valid measurement above the limit of quantitation without a protocol deviation with impact and for measurements that were above the limit of quantitation. (Age 2 to <6 years, 8.5 mg/kg has n = '0' since the values were below the limit of quantitation (BLQ).)
Measure: Mean (Standard Deviation); unit: hr*{Percent} inhibition P-selectin
Arm/Group | Age 12 to <18 Years, 5 mg/kg | Age 6 to <12 Years, 5 mg/kg | Age 6 to <12 Years, 8.5 mg/kg | Age 2 to <6 Years, 8.5 mg/kg
Number analyzed (Participants) | 11 | 12 | 13 | 0
hr*{Percent} inhibition P-selectin | 33700 (2440) | 34400 (3660) | 33200 (3410) |

5. Primary Outcome: Pharmacodynamics (PD) - P-selectin Inhibition Parameters for Crizanlizumab - Part A - AUCtau After Multiple Dose - Steady State
Description: The AUC of %inhibition calculated to the end of a dosing interval (tau) after multiple dose. AUCtau was calculated based on P-selectin inhibition curves.
Time Frame: Week 15 - Steady state
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr*{Percent} inhibition P-selectin
Arm/Group | Age 12 to <18 Years, 5 mg/kg | Age 6 to <12 Years, 5 mg/kg | Age 6 to <12 Years, 8.5 mg/kg | Age 2 to <6 Years, 8.5 mg/kg
Number analyzed (Participants) | 6 | 7 | 11 | 10
hr*{Percent} inhibition P-selectin | 66700 (9560) | 64800 (3550) | 68600 (9210) | 66300 (5710)

6. Primary Outcome: Frequency of Any Adverse Events (AEs) as a Measure of Safety and Tolerability
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a subject or clinical investigation subject
Time Frame: Adverse events are reported from the first dose of study treatment until end of study treatment Week 103 plus 105 days post-treatment follow-up, up to a maximum timeframe of approximately 2 years and 3.25 months.
Population: Safety analysis set - all treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Age 12 to <18 Years, 5 mg/kg | Age 6 to <12 Years, 5 mg/kg | Age 6 to <12 Years, 8.5 mg/kg | Age 2 to <6 Years, 8.5 mg/kg
Number analyzed (Participants) | 50 | 13 | 40 | 14
Participants
  Adverse events (AEs) | 47 | 13 | 38 | 14
  AEs -Treatment-related | 16 | 5 | 14 | 4
  Serious Adverse events (SAEs) | 18 | 9 | 20 | 12
  SAEs -Treatment-related | 1 | 1 | 2 | 1
  Fatal SAEs | 1 | 0 | 0 | 0
  Fatal SAEs-Treatment-related | 0 | 0 | 0 | 0
  AEs leading to dose interruption/reduction | 17 | 6 | 10 | 7
  AEs requiring additional therapy | 45 | 13 | 37 | 14

7. Secondary Outcome: Annualized Rate Vaso Occlusive Crisis (VOC) Events Leading to Healthcare Visit in Clinic / Emergency Room (ER) / Hospital
Description: VOC is defined as pain crises as well as other complicated crises, such as acute chest syndrome (ACS), priapism, and hepatic or splenic sequestration.
  The baseline annualized rate of VOC was defined as the number of VOCs leading to healthcare visit occurring within the last 12 months prior to screening until first dose.
  This annualized rate of VOC was calculated by multiplying the number of VOCs by 365 and dividing by the number of days in the observation period. (Parts A and B)
Time Frame: Baseline, Year 1 and Year 2
Population: Full analysis set - for treated participants with a valid measurement without a protocol deviation with impact who had VOC events leading to healthcare visit in clinic/ER/hospital.
Measure: Median (Full Range); unit: VOC events per year
Arm/Group | Age 12 to <18 Years, 5 mg/kg | Age 6 to <12 Years, 5 mg/kg | Age 6 to <12 Years, 8.5 mg/kg | Age 2 to <6 Years, 8.5 mg/kg
Number analyzed (Participants) | 50 | 13 | 40 | 14
VOC events per year
  Baseline annualized rate of VOC | 3.00 [1.0 to 26.0] | 1.00 [0.0 to 6.0] | 2.00 [1.0 to 13.0] | 1.00 [1.0 to 5.0]
  Annualized rate of VOC on treatment (up to Year 2) | 1.80 [0.0 to 14.5] | 0.79 [0.0 to 10.4] | 1.48 [0.0 to 8.7] | 1.22 [0.0 to 5.3]
  Annualized rate of VOC on treatment Year 1 (n=42,11,35,12): number analyzed (Participants) | 42 | 11 | 35 | 12
  Annualized rate of VOC on treatment Year 1 (n=42,11,35,12) | 2.00 [0.0 to 14.0] | 0.00 [0.0 to 4.0] | 1.00 [0.0 to 6.0] | 0.00 [0.0 to 3.0]
  Annualized rate of VOC on treatment Year 2 (n=32,10,27,10): number analyzed (Participants) | 32 | 10 | 27 | 10
  Annualized rate of VOC on treatment Year 2 (n=32,10,27,10) | 2.00 [0.0 to 8.0] | 0.00 [0.0 to 5.0] | 1.00 [0.0 to 9.0] | 2.00 [0.0 to 4.0]

8. Secondary Outcome: Annualized Rate Vaso Occlusive Crisis (VOC) Events Treated at Home (Based on Documentation by Health Care Provider Following Phone Contact With the Patient)
Description: VOC is defined as pain crises as well as other complicated crises, such as acute chest syndrome (ACS), priapism, and hepatic or splenic sequestration.
  This annualized rate of VOC was calculated by multiplying the number of VOCs by 365 and dividing by the number of days in the observation period. (Parts A and B)
Time Frame: Up to Year 2
Population: Full analysis set - for treated participants with a valid measurement without a protocol deviation with impact who had VOC events treated at home (based on documentation by health care provider following phone contact with the patient.
Measure: Median (Full Range); unit: VOC events per year
Arm/Group | Age 12 to <18 Years, 5 mg/kg | Age 6 to <12 Years, 5 mg/kg | Age 6 to <12 Years, 8.5 mg/kg | Age 2 to <6 Years, 8.5 mg/kg
Number analyzed (Participants) | 19 | 2 | 10 | 2
VOC events per year | 0.94 [0.5 to 3.9] | 2.71 [0.5 to 4.9] | 0.49 [0.49 to 3.0] | 0.73 [0.5 to 1.0]

9. Secondary Outcome: Annualized Rate Vaso Occlusive Crisis (VOC) Events Leading to Healthcare Visit - Uncomplicated Pain Crisis
Description: VOC is defined as pain crises as well as other complicated crises, such as acute chest syndrome (ACS), priapism, and hepatic or splenic sequestration.
  This annualized rate of VOC was calculated by multiplying the number of VOCs by 365 and dividing by the number of days in the observation period. (Parts A and B)
  Uncomplicated pain crisis is defined as an acute episode of pain with no known cause for pain other than a vaso-occlusive event; and requiring treatment with a parenteral or oral opioids or other parenteral analgesic; but is NOT classified as an acute chest syndrome, hepatic sequestration, splenic sequestration or priapism. The end of an uncomplicated pain crisis will be considered the resolution of acute pain, such that residual pain (or absence of any pain) is considered to be chronic, and the current pain medication regimen is considered to be for this chronic pain.
Time Frame: Up to Year 2
Population: Full analysis set - for treated participants with uncomplicated pain crisis without a protocol deviation with impact who had VOC events leading to healthcare visit - uncomplicated pain crisis.
Measure: Median (Full Range); unit: VOC events per year
Arm/Group | Age 12 to <18 Years, 5 mg/kg | Age 6 to <12 Years, 5 mg/kg | Age 6 to <12 Years, 8.5 mg/kg | Age 2 to <6 Years, 8.5 mg/kg
Number analyzed (Participants) | 50 | 12 | 38 | 14
VOC events per year | 1.79 [0.0 to 14.5] | 0.98 [0.0 to 10.4] | 1.47 [0.0 to 8.7] | 0.97 [0.0 to 5.3]

10. Secondary Outcome: Annualized Rate Vaso Occlusive Crisis (VOC) Events Leading to Healthcare Visit - Acute Chest Syndrome
Description: VOC is defined as pain crises as well as other complicated crises, such as acute chest syndrome (ACS), priapism, and hepatic or splenic sequestration.
  This annualized rate of VOC was calculated by multiplying the number of VOCs by 365 and dividing by the number of days in the observation period. (Parts A and B)
  Acute Chest Syndrome (ACS) is defined on the basis of the finding of a new pulmonary infiltrate involving at least one complete lung segment that was consistent with alveolar consolidation, but excluding atelectasis (as indicated by chest X-ray). At least one of the following additional signs or symptoms needs to be present as well: chest pain, a temperature of more than 38.5°C, tachypnea, wheezing or cough. ACS will be considered resolved when the patient is no longer hospitalized (unless for reason other than the ACS episode) and none of the additional signs or symptoms above are present (unless for reason other than the ACS).
Time Frame: Up to Year 2
Population: Full analysis set - for treated participants with acute chest syndrome without a protocol deviation with impact who had VOC events leading to healthcare visit - acute chest syndrome.
Measure: Median (Full Range); unit: VOC events per year
Arm/Group | Age 12 to <18 Years, 5 mg/kg | Age 6 to <12 Years, 5 mg/kg | Age 6 to <12 Years, 8.5 mg/kg | Age 2 to <6 Years, 8.5 mg/kg
Number analyzed (Participants) | 18 | 4 | 15 | 6
VOC events per year | 0.49 [0.0 to 3.7] | 0.64 [0.0 to 1.5] | 0.49 [0.0 to 1.0] | 0.49 [0.0 to 1.9]

11. Secondary Outcome: Annualized Rate Vaso Occlusive Crisis (VOC) Events Treated at Home (Based on Documentation by Health Care Provider Following Phone Contact With the Patient) - Hepatic Sequestration
Description: VOC is defined as pain crises as well as other complicated crises, such as acute chest syndrome (ACS), priapism, and hepatic or splenic sequestration.
  This annualized rate of VOC was calculated by multiplying the number of VOCs by 365 and dividing by the number of days in the observation period. (Parts A and B)
  Hepatic sequestration is defined on the basis of findings of right upper quadrant pain, an enlarged liver, and an acute decrease in hemoglobin concentration (e.g. a decrease in hemoglobin of ~ 2 g/dL). Acute hepatic sequestration will be considered resolved when right upper quadrant pain has returned to baseline (pre-event) levels and hemoglobin has been stable for 24 hrs.
  There were no patients with VOC events of hepatic sequestration treated at home. Therefore, there were no observations which met the report criteria.
Time Frame: Up to Year 2
Population: Full analysis set - for treated participants with hepatic sequestration without a protocol deviation with impact who had VOC events treated at home (based on documentation by health care provider following phone contact with the patient) - hepatic sequestration. There were no observations which met this criteria.
Arm/Group | Age 12 to <18 Years, 5 mg/kg | Age 6 to <12 Years, 5 mg/kg | Age 6 to <12 Years, 8.5 mg/kg | Age 2 to <6 Years, 8.5 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Annualized Rate Vaso Occlusive Crisis (VOC) Events Leading to Healthcare Visit - Splenic Sequestration
Description: VOC is defined as pain crises as well as other complicated crises, such as acute chest syndrome (ACS), priapism, and hepatic or splenic sequestration.
  This annualized rate of VOC was calculated by multiplying the number of VOCs by 365 and dividing by the number of days in the observation period. (Parts A and B)
  Splenic sequestration if defined on the basis of findings of left upper quadrant pain, an enlarged spleen, and an acute decrease in hemoglobin concentration (e.g., a decrease in hemoglobin of ~ 2 g/dL). Acute splenic sequestration will be considered resolved when left upper quadrant pain has returned to baseline (pre-event) levels and hemoglobin has been stable for 24 hrs.
Time Frame: Up to Year 2
Population: Full analysis set - for treated participants with splenic sequestration with a valid measurement and without a protocol deviation with impact who had VOC events leading to healthcare visit - splenic sequestration. (No patients in the 4th group met this criteria.)
Measure: Median (Full Range); unit: VOC events per year
Arm/Group | Age 12 to <18 Years, 5 mg/kg | Age 6 to <12 Years, 5 mg/kg | Age 6 to <12 Years, 8.5 mg/kg | Age 2 to <6 Years, 8.5 mg/kg
Number analyzed (Participants) | 3 | 1 | 1 | 0
VOC events per year | 0.00 [0.0 to 0.5] | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0] |

13. Secondary Outcome: Annualized Rate Vaso Occlusive Crisis (VOC) Events Leading to Healthcare Visit - Priapism
Description: VOC is defined as pain crises as well as other complicated crises, such as acute chest syndrome (ACS), priapism, and hepatic or splenic sequestration.
  This annualized rate of VOC was calculated by multiplying the number of VOCs by 365 and dividing by the number of days in the observation period. (Parts A and B)
  Priapism is defined as an unwanted or painful penile erection lasting at least 30 minutes. The end of an acute priapism event will be when the unwanted erection has resolved for at least 2 hours.
Time Frame: Up to Year 2
Population: Full analysis set - for treated participants with priapism and with a valid measurement above the limit of quantitation without a protocol deviation with impact who had VOC events leading to healthcare visit - priapism. (No patients in the 1st and 4th group met this criteria.)
Measure: Median (Full Range); unit: VOC events per year
Arm/Group | Age 12 to <18 Years, 5 mg/kg | Age 6 to <12 Years, 5 mg/kg | Age 6 to <12 Years, 8.5 mg/kg | Age 2 to <6 Years, 8.5 mg/kg
Number analyzed (Participants) | 0 | 1 | 1 | 0
VOC events per year |  | 0.49 [0.49 to 0.49] | 0.00 [0.0 to 0.0] |

14. Secondary Outcome: Annualized Rate of Hospitalizations and Emergency Room (ER) Visits (VOC-related)
Description: VOC is defined as pain crises as well as other complicated crises, such as acute chest syndrome (ACS), priapism, and hepatic or splenic sequestration.
  This rate was calculated by multiplying the number of hospitalizations and ER visits (VOC-related) by 365 and dividing by the number of days in the observation period.
  Units would be something like: hospitalizations and ER visits per year. (Parts A and B)
Time Frame: Up to Year 2
Population: Full analysis set - for treated participants with a valid measurement without a protocol deviation with impact who had hospitalizations and ER visits (VOC-related).
Measure: Median (Full Range); unit: hospitalizations and ER visits per year
Arm/Group | Age 12 to <18 Years, 5 mg/kg | Age 6 to <12 Years, 5 mg/kg | Age 6 to <12 Years, 8.5 mg/kg | Age 2 to <6 Years, 8.5 mg/kg
Number analyzed (Participants) | 50 | 13 | 40 | 14
hospitalizations and ER visits per year
  Annualized rate of hospitalizations and ER visits (up to Year 2) | 1.78 [0.0 to 13.5] | 0.50 [0.0 to 10.4] | 1.01 [0.0 to 9.6] | 0.74 [0.0 to 5.3]
  Annualized rate of hospitalizations and ER visits Year 1 (n=42,11,35,12): number analyzed (Participants) | 42 | 11 | 35 | 12
  Annualized rate of hospitalizations and ER visits Year 1 (n=42,11,35,12) | 2.00 [0.0 to 14.0] | 0.00 [0.0 to 5.0] | 1.00 [0.0 to 6.0] | 0.00 [0.0 to 3.0]
  Annualized rate of hospitalizations and ER visits Year 2 (n=32,10,27,10): number analyzed (Participants) | 32 | 10 | 27 | 10
  Annualized rate of hospitalizations and ER visits Year 2 (n=32,10,27,10) | 2.00 [0.0 to 9.0] | 0.00 [0.0 to 5.0] | 1.00 [0.0 to 10.0] | 1.00 [0.0 to 3.0]

15. Secondary Outcome: Annualized Rate of Hospitalizations and Emergency Room (ER) Visits (Total)
Description: VOC is defined as pain crises as well as other complicated crises, such as acute chest syndrome (ACS), priapism, and hepatic or splenic sequestration.
  The baseline annualized rate of VOC was defined as the number of VOCs leading to healthcare visit occurring within the last 12 months prior to screening until first dose.
  This rate was calculated by multiplying the number of hospitalizations and ER visits (VOC-related) by 365 and dividing by the number of days in the observation period.
  Units would be something like: hospitalizations and ER visits per year. (Parts A and B)
Time Frame: Up to Year 2
Population: Full analysis set - for treated participants with a valid measurement without a protocol deviation with impact who had hospitalizations and ER visits.
Measure: Median (Full Range); unit: hospitalizations and ER visits per year
Arm/Group | Age 12 to <18 Years, 5 mg/kg | Age 6 to <12 Years, 5 mg/kg | Age 6 to <12 Years, 8.5 mg/kg | Age 2 to <6 Years, 8.5 mg/kg
Number analyzed (Participants) | 50 | 13 | 40 | 14
hospitalizations and ER visits per year
  Annualized rate of hospitalizations and ER visits (up to Year 2) | 2.68 [0.0 to 15.5] | 1.46 [0.0 to 11.4] | 1.59 [0.0 to 11.7] | 1.74 [0.0 to 7.7]
  Annualized rate of hospitalizations and ER visits Year 1 (n=42,11,35,12): number analyzed (Participants) | 42 | 11 | 35 | 12
  Annualized rate of hospitalizations and ER visits Year 1 (n=42,11,35,12) | 2.00 [0.0 to 16.0] | 1.00 [0.0 to 5.0] | 2.00 [0.0 to 7.0] | 2.00 [0.0 to 8.0]
  Annualized rate of hospitalizations and ER visits Year 2 (n=32,10,27,10): number analyzed (Participants) | 32 | 10 | 27 | 10
  Annualized rate of hospitalizations and ER visits Year 2 (n=32,10,27,10) | 2.50 [0.0 to 10.0] | 1.00 [0.0 to 8.0] | 1.00 [0.0 to 10.0] | 2.00 [0.0 to 4.0]

16. Secondary Outcome: Annualized Days of Emergency Room (ER) / Hospitalization (Both Overall and VOC-related)
Description: VOC is defined as pain crises as well as other complicated crises, such as acute chest syndrome (ACS), priapism, and hepatic or splenic sequestration.
  The baseline annualized rate of VOC was defined as the number of VOCs leading to healthcare visit occurring within the last 12 months prior to screening until first dose.
  This rate was calculated by multiplying the number of days of ER/hospitalizations (both overall and VOC-related) by 365 and dividing by the number of days in the observation period. (Parts A and B)
Time Frame: Years 1 and 2
Population: Full analysis set - for treated participants with a valid measurement without a protocol deviation with impact who had ER/hospitalizations.
Measure: Median (Full Range); unit: Days per year
Arm/Group | Age 12 to <18 Years, 5 mg/kg | Age 6 to <12 Years, 5 mg/kg | Age 6 to <12 Years, 8.5 mg/kg | Age 2 to <6 Years, 8.5 mg/kg
Number analyzed (Participants) | 50 | 13 | 40 | 14
Days per year
  Annualized days of ER/Hospitalization on treatment - VOC related (up to Year 2) | 6.74 [0.0 to 87.0] | 0.98 [0.0 to 59.2] | 5.36 [0.0 to 40.0] | 2.20 [0.0 to 42.7]
  Annualized days of ER/Hospitalization on treatment - Total (up to Year 2) | 12.37 [0.0 to 87.0] | 5.41 [0.0 to 59.2] | 9.03 [0.0 to 57.5] | 10.48 [0.0 to 42.7]
  Annualized days of ER/Hospitalization Year 1 - VOC related (n=42,11,12, 12): number analyzed (Participants) | 42 | 11 | 12 | 12
  Annualized days of ER/Hospitalization Year 1 - VOC related (n=42,11,12, 12) | 7.00 [0.0 to 60.3] | 0.00 [0.0 to 23.0] | 5.00 [0.0 to 37.0] | 0.00 [0.0 to 29.0]
  Annualized days of ER/Hospitalization Year 1 - Total (n=42,11,12, 12): number analyzed (Participants) | 42 | 11 | 12 | 12
  Annualized days of ER/Hospitalization Year 1 - Total (n=42,11,12, 12) | 7.00 [0.0 to 60.3] | 2.00 [0.0 to 24.0] | 11.00 [0.0 to 37.0] | 6.50 [0.0 to 34.0]
  Annualized days of ER/Hospitalization Year 2 - VOC related (n=32,10,11, 10): number analyzed (Participants) | 32 | 10 | 11 | 10
  Annualized days of ER/Hospitalization Year 2 - VOC related (n=32,10,11, 10) | 10.50 [0.0 to 71.0] | 0.00 [0.0 to 48.0] | 2.00 [0.0 to 40.0] | 3.00 [0.0 to 19.0]
  Annualized days of ER/Hospitalization Year 2 - Total (n=32,10,11, 10): number analyzed (Participants) | 32 | 10 | 11 | 10
  Annualized days of ER/Hospitalization Year 2 - Total (n=32,10,11, 10) | 13.00 [0.0 to 71.0] | 2.00 [0.0 to 64.0] | 3.00 [0.0 to 40.0] | 10.50 [0.0 to 37.0]

17. Secondary Outcome: Annualized Rate of Dactylitis Events
Description: Dactylitis, also known as 'hand-foot syndrome', is a complication of acute vaso-occlusive disease characterized by pain and edema of the digits as well as the dorsum of the hands or feet, or both simultaneously, often accompanied by increased local temperature and erythema.
  There were no patients with dactylitis events. Therefore, there were no observations which met the report criteria.
Time Frame: On Treatment, up to Year 2
Population: Safety analysis set - all treated participants who had dactylitis events. There were no observations which met the report criteria.
Arm/Group | Age 12 to <18 Years, 5 mg/kg | Age 6 to <12 Years, 5 mg/kg | Age 6 to <12 Years, 8.5 mg/kg | Age 2 to <6 Years, 8.5 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0

18. Secondary Outcome: Absolute Change From Baseline in Hemoglobin
Description: Hemoglobin is a protein that carries oxygen through the body. It attaches to red blood cells, delivers oxygen throughout the body, and transports carbon dioxide back to the lungs. In sickle cell disease, red blood cells are crescent or sickle-shaped due to a genetic mutation, and those sickled red blood cells can clog blood flow, causing debilitating pain and even organ damage.
Time Frame: Baseline, Week 27, Year 2
Population: Safety analysis set - for treated participants with a valid measurement without a protocol deviation with impact.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Age 12 to <18 Years, 5 mg/kg | Age 6 to <12 Years, 5 mg/kg | Age 6 to <12 Years, 8.5 mg/kg | Age 2 to <6 Years, 8.5 mg/kg
Number analyzed (Participants) | 39 | 9 | 36 | 11
g/L
  Week 27 | -1.26 (11.472) | 2.33 (6.856) | -0.33 (7.015) | 1.55 (9.905)
  End Of Treatment / Year 2 (n=24,6,11,2): number analyzed (Participants) | 24 | 6 | 11 | 2
  End Of Treatment / Year 2 (n=24,6,11,2) | -5.38 (11.088) | 2.33 (7.941) | -1.18 (11.677) | 15.00 (1.414)

19. Secondary Outcome: Immunogenicity: Measurement of Anti-drug Antibodies (ADA) to Crizanlizumab
Description: Anti-drug antibodies (ADA) are antibodies elicited from therapeutics and they are used to measure immunogenicity.
Time Frame: up to Year 2
Population: Full analysis set - for treated participants with a valid measurement without a protocol deviation with impact.
Measure: Count of Participants; unit: Participants
Arm/Group | Age 12 to <18 Years, 5 mg/kg | Age 6 to <12 Years, 5 mg/kg | Age 6 to <12 Years, 8.5 mg/kg | Age 2 to <6 Years, 8.5 mg/kg
Number analyzed (Participants) | 50 | 13 | 39 | 14
Participants
  Baseline - Negative | 50 | 13 | 39 | 14
  Baseline - Positive | 0 | 0 | 0 | 0
  Baseline - Missing | 0 | 0 | 1 | 0
  Post-baseline - Any positive | 0 | 1 | 1 | 0
  Post-baseline - only last sample positive | 0 | 0 | 0 | 0

20. Secondary Outcome: Notable On-treatment Findings From the Electrocardiogram (ECG) Assessments
Description: QTcF = QT interval corrected by Fridericia's formula QTcB = Corrected QT interval Bazett's Formula QT = QT interval PR = PR interval QRS = QRS interval RR = RR interval HR = heart rate
Time Frame: Baseline, up to Year 2
Population: Safety analysis set - for treated participants with a valid measurement without a protocol deviation with impact
Measure: Count of Participants; unit: Participants
Arm/Group | Age 12 to <18 Years, 5 mg/kg | Age 6 to <12 Years, 5 mg/kg | Age 6 to <12 Years, 8.5 mg/kg | Age 2 to <6 Years, 8.5 mg/kg
Number analyzed (Participants) | 49 | 13 | 40 | 13
Participants
  QTcF (ms)-Increase >30 to <=60 ms (n=49,13,37,12): number analyzed (Participants) | 49 | 13 | 37 | 12
  QTcF (ms)-Increase >30 to <=60 ms (n=49,13,37,12) | 1 | 1 | 2 | 1
  QTcF (ms)- Increase >60 ms (n=49,13,37,12): number analyzed (Participants) | 49 | 13 | 37 | 12
  QTcF (ms)- Increase >60 ms (n=49,13,37,12) | 0 | 0 | 0 | 0
  QTcF (ms)- New >450 to <=480 ms (n=49,13,40,13) | 3 | 0 | 0 | 0
  QTcF (ms)- New >480 to <=500 ms (n=49,13,40,13) | 0 | 0 | 1 | 0
  QTcF (ms)-New >500 ms (n=49,13,40,13) | 0 | 0 | 0 | 0
  QTcB (ms)-Increase >30 to <=60 ms (n=49,13,37,12): number analyzed (Participants) | 49 | 13 | 37 | 12
  QTcB (ms)-Increase >30 to <=60 ms (n=49,13,37,12) | 12 | 3 | 7 | 1
  QTcB (ms)-Increase >60 ms (n=49,13,37,12): number analyzed (Participants) | 49 | 13 | 37 | 12
  QTcB (ms)-Increase >60 ms (n=49,13,37,12) | 0 | 0 | 0 | 0
  QTcB (ms)-New >450 to <=480 ms (n=40,12,35,13): number analyzed (Participants) | 40 | 12 | 35 | 13
  QTcB (ms)-New >450 to <=480 ms (n=40,12,35,13) | 10 | 2 | 14 | 6
  QTcB (ms)-New >480 to <=500 ms (n=49,13,40,13) | 3 | 0 | 1 | 0
  QTcB (ms)-New >500 ms (n=49,13,40,13) | 0 | 0 | 0 | 0
  QT (ms)-Increase >30 to <=60 ms (n=49,13,37,12): number analyzed (Participants) | 49 | 13 | 37 | 12
  QT (ms)-Increase >30 to <=60 ms (n=49,13,37,12) | 13 | 5 | 17 | 3
  QT (ms)-Increase >60 ms (n=49,13,37,12): number analyzed (Participants) | 49 | 13 | 37 | 12
  QT (ms)-Increase >60 ms (n=49,13,37,12) | 2 | 0 | 2 | 0
  QT (ms)-New >450 to <=480 ms (n=49,13,40,13) | 0 | 0 | 0 | 0
  QT (ms)-New >480 to <=500 ms (n=49,13,40,13) | 0 | 0 | 0 | 0
  QT (ms)-New >500 ms (n=49,13,40,13) | 0 | 0 | 0 | 0
  PR (ms)-Increase >25% and PR >200 ms (n=48,13,37,12): number analyzed (Participants) | 48 | 13 | 37 | 12
  PR (ms)-Increase >25% and PR >200 ms (n=48,13,37,12) | 0 | 0 | 0 | 0
  PR (ms)-New PR >200 ms (n=48,13,40,13): number analyzed (Participants) | 48 | 13 | 40 | 13
  PR (ms)-New PR >200 ms (n=48,13,40,13) | 2 | 0 | 0 | 0
  QRS (ms)- Increase >25% and QRS >120 ms (n=49,13,37,12): number analyzed (Participants) | 49 | 13 | 37 | 12
  QRS (ms)- Increase >25% and QRS >120 ms (n=49,13,37,12) | 0 | 0 | 0 | 0
  QRS (ms)-New QRS >120 ms (n=49,13,40,13) | 0 | 0 | 0 | 0
  RR (ms)-Increase >25% and RR >1200 ms (n=49,13,37,12): number analyzed (Participants) | 49 | 13 | 37 | 12
  RR (ms)-Increase >25% and RR >1200 ms (n=49,13,37,12) | 1 | 0 | 0 | 0
  RR (ms)-Decrease >25% and RR <600 ms (n=49,12,34,7): number analyzed (Participants) | 49 | 12 | 34 | 7
  RR (ms)-Decrease >25% and RR <600 ms (n=49,12,34,7) | 0 | 1 | 2 | 0
  HR (bpm)-Increase >25% and HR >100 bpm (n=49,12,34,7): number analyzed (Participants) | 49 | 12 | 34 | 7
  HR (bpm)-Increase >25% and HR >100 bpm (n=49,12,34,7) | 1 | 1 | 3 | 0
  HR (bpm)-Decrease >25% and HR <50 bpm (n=49,13,37,12): number analyzed (Participants) | 49 | 13 | 37 | 12
  HR (bpm)-Decrease >25% and HR <50 bpm (n=49,13,37,12) | 0 | 0 | 0 | 0

21. Secondary Outcome: Growth and Sexual Maturation Assessments (Tanner Stage) - Abnormalities - for Female Participants at Risk of Delayed Puberty at Start Date of Study Treatment
Description: As assessed per Tanner criteria.
  The number of Participants Analyzed row refer to participants who have not started puberty and have not had delayed puberty prior to start date of study treatment.
  Delayed puberty in females is defined as failure to attain Tanner Stage 2 (for both breast development and pubic hair) by age 13, or absence of menarche by age 15 or within 5 years of attainment of Tanner Stage 2.
Time Frame: Week 51
Population: Full analysis set - only for participants at risk of delayed puberty, (i.e., excludes participants who already reached puberty at study start.)
Measure: Count of Participants; unit: Participants
Arm/Group | Age 12 to <18 Years, 5 mg/kg | Age 6 to <12 Years, 5 mg/kg | Age 6 to <12 Years, 8.5 mg/kg | Age 2 to <6 Years, 8.5 mg/kg
Number analyzed (Participants) | 0 | 3 | 12 | 5
Participants
  Delayed puberty = yes |  | 0 | 0 | 0
  Delayed puberty = no |  | 0 | 0 | 0
  Delayed puberty = unknown (i.e., not applicable because pt not yet in age range for puberty) |  | 3 | 12 | 5

22. Secondary Outcome: Growth and Sexual Maturation Assessments (Tanner Stage) - Abnormalities - for Male Participants at Risk of Delayed Puberty at Start Date of Study Treatment
Description: As assessed per Tanner criteria.
  The number of Participants Analyzed row refer to participants who have not started puberty and have not had delayed puberty prior to start date of study treatment.
  Delayed puberty in males is defined as failure to attain Tanner Stage 2 (for both genitalia and pubic hair) by age 14.
Time Frame: Week 51
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Age 12 to <18 Years, 5 mg/kg | Age 6 to <12 Years, 5 mg/kg | Age 6 to <12 Years, 8.5 mg/kg | Age 2 to <6 Years, 8.5 mg/kg
Number analyzed (Participants) | 4 | 7 | 18 | 9
Participants
  Delayed puberty = yes | 0 | 0 | 0 | 0
  Delayed puberty = no | 4 | 0 | 0 | 0
  Delayed puberty = unknown (i.e., not applicable because pt not yet in age range for puberty) | 0 | 7 | 18 | 9

23. Secondary Outcome: PK Pre-dose Concentrations of Crizanlizumab Prior to Each Study Drug Dose - Part A
Time Frame: Week 3, Week 7, Week 11, Week 15, Week 19, Week 23, Week 27, Week 31, Week 35, Week 39, Week 43, Week 47 and Week 51 (Day 1, 0 hr (pre-dose))
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Age 12 to <18 Years, 5 mg/kg | Age 6 to <12 Years, 5 mg/kg | Age 6 to <12 Years, 8.5 mg/kg | Age 2 to <6 Years, 8.5 mg/kg
Number analyzed (Participants) | 11 | 12 | 13 | 12
µg/mL
  Week 3 Day 1, 0 hr (pre-dose) (n=11,12,13,10): number analyzed (Participants) | 11 | 12 | 13 | 10
  Week 3 Day 1, 0 hr (pre-dose) (n=11,12,13,10) | 16.8 (4.40) | 14.1 (5.61) | 30.1 (6.17) | 19.8 (5.62)
  Week 7 Day 1, 0 hr (pre-dose) (n=9,12,12,12): number analyzed (Participants) | 9 | 12 | 12 | 12
  Week 7 Day 1, 0 hr (pre-dose) (n=9,12,12,12) | 10.7 (3.30) | 8.70 (5.32) | 22.1 (8.09) | 13.4 (3.21)
  Week 11 Day 1, 0 hr (pre-dose) (n=9,11,12,11): number analyzed (Participants) | 9 | 11 | 12 | 11
  Week 11 Day 1, 0 hr (pre-dose) (n=9,11,12,11) | 10.2 (4.92) | 6.02 (4.43) | 20.1 (9.36) | 11.0 (3.80)
  Week 15 Day 1, 0 hr (pre-dose) (n=7,9,11,12): number analyzed (Participants) | 7 | 9 | 11 | 12
  Week 15 Day 1, 0 hr (pre-dose) (n=7,9,11,12) | 9.42 (6.47) | 8.45 (2.93) | 20.4 (7.22) | 10.3 (5.84)
  Week 19 Day 1, 0 hr (pre-dose) (n=6,9,12,11): number analyzed (Participants) | 6 | 9 | 12 | 11
  Week 19 Day 1, 0 hr (pre-dose) (n=6,9,12,11) | 6.77 (4.53) | 7.75 (4.92) | 18.8 (5.28) | 10.2 (5.93)
  Week 23 Day 1, 0 hr (pre-dose) (n=9,12,12,10): number analyzed (Participants) | 9 | 12 | 12 | 10
  Week 23 Day 1, 0 hr (pre-dose) (n=9,12,12,10) | 6.17 (3.92) | 7.15 (5.23) | 20.0 (6.74) | 10.6 (5.24)
  Week 27 Day 1, 0 hr (pre-dose) (n=9,10,12,10): number analyzed (Participants) | 9 | 10 | 12 | 10
  Week 27 Day 1, 0 hr (pre-dose) (n=9,10,12,10) | 8.05 (5.32) | 7.70 (5.93) | 22.4 (8.71) | 11.8 (9.30)
  Week 31 Day 1, 0 hr (pre-dose) (n=6,10,11,10): number analyzed (Participants) | 6 | 10 | 11 | 10
  Week 31 Day 1, 0 hr (pre-dose) (n=6,10,11,10) | 9.46 (4.34) | 8.57 (6.17) | 19.3 (6.36) | 9.68 (8.29)
  Week 35 Day 1, 0 hr (pre-dose) (n=5,11,10,9): number analyzed (Participants) | 5 | 11 | 10 | 9
  Week 35 Day 1, 0 hr (pre-dose) (n=5,11,10,9) | 12.0 (6.04) | 6.88 (3.04) | 17.9 (8.03) | 8.43 (6.78)
  Week 39 Day 1, 0 hr (pre-dose) (n=7,11,10,11): number analyzed (Participants) | 7 | 11 | 10 | 11
  Week 39 Day 1, 0 hr (pre-dose) (n=7,11,10,11) | 4.93 (3.00) | 7.04 (5.75) | 19.9 (5.21) | 12.8 (7.98)
  Week 43 Day 1, 0 hr (pre-dose) (n=8,10,11,8): number analyzed (Participants) | 8 | 10 | 11 | 8
  Week 43 Day 1, 0 hr (pre-dose) (n=8,10,11,8) | 9.23 (4.73) | 7.45 (5.66) | 18.0 (8.07) | 12.8 (4.95)
  Week 47 Day 1, 0 hr (pre-dose) (n=8,8,10,10): number analyzed (Participants) | 8 | 8 | 10 | 10
  Week 47 Day 1, 0 hr (pre-dose) (n=8,8,10,10) | 7.32 (3.84) | 10.4 (7.29) | 14.6 (8.22) | 10.5 (9.26)
  Week 51 Day 1, 0 hr (pre-dose) (n=5,9,10,8): number analyzed (Participants) | 5 | 9 | 10 | 8
  Week 51 Day 1, 0 hr (pre-dose) (n=5,9,10,8) | 9.78 (6.61) | 9.44 (8.22) | 12.8 (10.6) | 10.3 (3.21)

24. Secondary Outcome: PK Pre-dose Concentrations of Crizanlizumab Prior to Each Study Drug Dose - Parts A and B
Time Frame: Week 3, Week 7, Week 11, Week 15, Week 19, Week 23, Week 27, Week 31, Week 35, Week 39, Week 43, Week 47 and Week 51 (0 hr (pre-dose))
Population: Pharmacokinetic analysis set 2 - for treated participants with a valid measurement without a protocol deviation with impact.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Age 12 to <18 Years, 5 mg/kg | Age 6 to <12 Years, 5 mg/kg | Age 6 to <12 Years, 8.5 mg/kg | Age 2 to <6 Years, 8.5 mg/kg
Number analyzed (Participants) | 45 | 12 | 36 | 13
µg/mL
  Week 3 Day 1, 0 hr (pre-dose) (n=45,12,36,11): number analyzed (Participants) | 45 | 12 | 36 | 11
  Week 3 Day 1, 0 hr (pre-dose) (n=45,12,36,11) | 16.6 (4.40) | 14.1 (5.61) | 23.6 (7.54) | 20.0 (5.37)
  Week 7 Day 1, 0 hr (pre-dose) (n=44,12,35,13): number analyzed (Participants) | 44 | 12 | 35 | 13
  Week 7 Day 1, 0 hr (pre-dose) (n=44,12,35,13) | 10.3 (5.49) | 8.70 (5.32) | 16.3 (7.50) | 14.4 (4.57)
  Week 11 Day 1, 0 hr (pre-dose)(n=45,11,33,11): number analyzed (Participants) | 45 | 11 | 33 | 11
  Week 11 Day 1, 0 hr (pre-dose)(n=45,11,33,11) | 9.18 (5.57) | 6.02 (4.43) | 15.3 (7.78) | 11.0 (3.80)
  Week 15 Day 1, 0 hr (pre-dose) (n=39,9,33,12): number analyzed (Participants) | 39 | 9 | 33 | 12
  Week 15 Day 1, 0 hr (pre-dose) (n=39,9,33,12) | 8.65 (5.73) | 8.45 (2.93) | 16.7 (7.34) | 10.3 (5.84)
  Week 19 Day 1, 0 hr (pre-dose) (n=38,9,35,11): number analyzed (Participants) | 38 | 9 | 35 | 11
  Week 19 Day 1, 0 hr (pre-dose) (n=38,9,35,11) | 8.13 (5.65) | 7.75 (4.92) | 17.5 (5.93) | 10.2 (5.93)
  Week 23 Day 1, 0 hr (pre-dose) (n=43,12,35,10): number analyzed (Participants) | 43 | 12 | 35 | 10
  Week 23 Day 1, 0 hr (pre-dose) (n=43,12,35,10) | 7.09 (4.45) | 7.15 (5.23) | 16.6 (6.90) | 10.6 (5.24)
  Week 27 Day 1, 0 hr (pre-dose) (n=40,10,34,10): number analyzed (Participants) | 40 | 10 | 34 | 10
  Week 27 Day 1, 0 hr (pre-dose) (n=40,10,34,10) | 7.07 (4.26) | 7.70 (5.93) | 16.5 (8.45) | 11.8 (9.30)
  Week 31 Day 1, 0 hr (pre-dose) (n=39,10,35,10): number analyzed (Participants) | 39 | 10 | 35 | 10
  Week 31 Day 1, 0 hr (pre-dose) (n=39,10,35,10) | 7.30 (4.80) | 8.57 (6.17) | 16.1 (7.57) | 9.68 (8.29)
  Week 35 Day 1, 0 hr (pre-dose) (n=35,11,32,10): number analyzed (Participants) | 35 | 11 | 32 | 10
  Week 35 Day 1, 0 hr (pre-dose) (n=35,11,32,10) | 8.96 (4.94) | 6.88 (3.04) | 13.6 (7.75) | 10.0 (8.11)
  Week 39 Day 1, 0 hr (pre-dose) (n=38,11,35,12): number analyzed (Participants) | 38 | 11 | 35 | 12
  Week 39 Day 1, 0 hr (pre-dose) (n=38,11,35,12) | 7.69 (5.46) | 7.04 (5.75) | 14.2 (7.79) | 13.4 (7.89)
  Week 43 Day 1, 0 hr (pre-dose) (n=35,10,34,9): number analyzed (Participants) | 35 | 10 | 34 | 9
  Week 43 Day 1, 0 hr (pre-dose) (n=35,10,34,9) | 8.68 (4.50) | 7.45 (5.66) | 14.8 (6.94) | 13.6 (5.15)
  Week 47 Day 1, 0 hr (pre-dose): number analyzed (Participants) | 38 | 8 | 34 | 10
  Week 47 Day 1, 0 hr (pre-dose) | 8.99 (5.76) | 10.4 (7.29) | 13.8 (6.80) | 10.5 (9.26)
  Week 51 Day 1, 0 hr (pre-dose): number analyzed (Participants) | 37 | 9 | 28 | 9
  Week 51 Day 1, 0 hr (pre-dose) | 8.48 (5.48) | 9.44 (8.22) | 13.4 (7.90) | 11.6 (4.90)

25. Secondary Outcome: Percent P-selectin Inhibition of Crizanlizumab Prior to Dosing - Part A
Description: A PD marker of crizanlizumab is the ex vivo P-selectin inhibition measured by a surface plasmon resonance assay using human serum samples. Crizanlizumab in serum samples binds to spiked Psel-Ig (P-selectin coupled to Ig) and inhibits its binding to a PSGL1 peptide.
Time Frame: Weeks 3, 7, 11,15, 19, 23, 27, 31, 35, 39, 43,47,51 (Day 1, 0 hr (pre-dose))
Population: Pharmacodynamic analysis set 1 - for treated participants with a valid measurement without a protocol deviation with impact.
Measure: Mean (Standard Deviation); unit: % inhibition P-selectin
Arm/Group | Age 12 to <18 Years, 5 mg/kg | Age 6 to <12 Years, 5 mg/kg | Age 6 to <12 Years, 8.5 mg/kg | Age 2 to <6 Years, 8.5 mg/kg
Number analyzed (Participants) | 11 | 12 | 13 | 10
% inhibition P-selectin
  Week 3 Day 1, 0 hr (pre-dose) (n=11,12,13,9): number analyzed (Participants) | 11 | 12 | 13 | 9
  Week 3 Day 1, 0 hr (pre-dose) (n=11,12,13,9) | 100 (0.0924) | 97.9 (2.97) | 99.1 (1.41) | 98.6 (2.54)
  Week 7 Day 1, 0 hr (pre-dose) (n=9,11,12,10): number analyzed (Participants) | 9 | 11 | 12 | 10
  Week 7 Day 1, 0 hr (pre-dose) (n=9,11,12,10) | 99.0 (1.61) | 94.2 (12.2) | 98.5 (3.48) | 98.9 (1.91)
  Week 11 Day 1, 0 hr (pre-dose) (n=9,9,12,9): number analyzed (Participants) | 9 | 9 | 12 | 9
  Week 11 Day 1, 0 hr (pre-dose) (n=9,9,12,9) | 97.7 (4.56) | 80.8 (32.4) | 98.5 (2.93) | 98.4 (2.50)
  Week 15 Day 1, 0 hr (pre-dose) (n=6,8,11,10): number analyzed (Participants) | 6 | 8 | 11 | 10
  Week 15 Day 1, 0 hr (pre-dose) (n=6,8,11,10) | 96.6 (8.04) | 99.8 (0.422) | 99.2 (1.86) | 91.7 (19.8)
  Week 19 Day 1, 0 hr (pre-dose) (n=6,9,12,10): number analyzed (Participants) | 6 | 9 | 12 | 10
  Week 19 Day 1, 0 hr (pre-dose) (n=6,9,12,10) | 88.6 (20.6) | 83.5 (34.8) | 99.2 (1.54) | 96.7 (5.51)
  Week 23 Day 1, 0 hr (pre-dose) (n=9,10,11,9): number analyzed (Participants) | 9 | 10 | 11 | 9
  Week 23 Day 1, 0 hr (pre-dose) (n=9,10,11,9) | 83.8 (28.9) | 91.2 (14.0) | 99.5 (1.24) | 92.2 (15.7)
  Week 27 Day 1, 0 hr (pre-dose) (n=9,9,11,8): number analyzed (Participants) | 9 | 9 | 11 | 8
  Week 27 Day 1, 0 hr (pre-dose) (n=9,9,11,8) | 88.0 (25.0) | 90.8 (20.4) | 99.4 (1.36) | 85.4 (19.1)
  Week 31 Day 1, 0 hr (pre-dose) (n=6,9,9,9): number analyzed (Participants) | 6 | 9 | 9 | 9
  Week 31 Day 1, 0 hr (pre-dose) (n=6,9,9,9) | 97.8 (2.83) | 88.9 (21.0) | 99.6 (1.30) | 75.5 (37.9)
  Week 35 Day 1, 0 hr (pre-dose) (n=5,10,8,9): number analyzed (Participants) | 5 | 10 | 8 | 9
  Week 35 Day 1, 0 hr (pre-dose) (n=5,10,8,9) | 97.2 (6.04) | 92.3 (10.6) | 97.9 (3.81) | 67.4 (42.1)
  Week 39 Day 1, 0 hr (pre-dose) (n=7,7,8,9): number analyzed (Participants) | 7 | 7 | 8 | 9
  Week 39 Day 1, 0 hr (pre-dose) (n=7,7,8,9) | 80.8 (28.0) | 88.6 (25.3) | 99.1 (2.01) | 87.6 (19.2)
  Week 43 Day 1, 0 hr (pre-dose) (n=8,3,9,6): number analyzed (Participants) | 8 | 3 | 9 | 6
  Week 43 Day 1, 0 hr (pre-dose) (n=8,3,9,6) | 96.7 (4.19) | 99.0 (1.67) | 98.8 (2.14) | 98.8 (2.37)
  Week 47 Day 1, 0 hr (pre-dose) (n=8,2,8,8): number analyzed (Participants) | 8 | 2 | 8 | 8
  Week 47 Day 1, 0 hr (pre-dose) (n=8,2,8,8) | 87.1 (30.5) | 98.8 (1.77) | 98.1 (3.73) | 69.8 (44.0)
  Week 51 Day 1, 0 hr (pre-dose) (n=5,3,8,7): number analyzed (Participants) | 5 | 3 | 8 | 7
  Week 51 Day 1, 0 hr (pre-dose) (n=5,3,8,7) | 80.9 (34.0) | 95.4 (4.24) | 98.9 (1.86) | 92.1 (13.0)

26. Secondary Outcome: Percent P-selectin Inhibition of Crizanlizumab Prior to Dosing - Part A and B
Description: as for outcome 25
Time Frame: Weeks 3, 7, 11,15, 19, 23, 27, 31, 35, 39, 43,47,51 (Day 1, 0 hr (pre-dose))
Population: Pharmacodynamic analysis set 2 - for treated participants with a valid measurement without a protocol deviation with impact.
Measure: Mean (Standard Deviation); unit: % inhibition P-selectin
Arm/Group | Age 12 to <18 Years, 5 mg/kg | Age 6 to <12 Years, 5 mg/kg | Age 6 to <12 Years, 8.5 mg/kg | Age 2 to <6 Years, 8.5 mg/kg
Number analyzed (Participants) | 42 | 12 | 36 | 12
% inhibition P-selectin
  Week 3 Day 1, 0 hr (pre-dose) (n=42,12,36,11): number analyzed (Participants) | 42 | 12 | 36 | 11
  Week 3 Day 1, 0 hr (pre-dose) (n=42,12,36,11) | 99.3 (2.14) | 97.9 (2.97) | 98.3 (3.74) | 97.6 (3.71)
  Week 7 Day 1, 0 hr (pre-dose) (n=41,12,35,12): number analyzed (Participants) | 41 | 12 | 35 | 12
  Week 7 Day 1, 0 hr (pre-dose) (n=41,12,35,12) | 93.7 (17.0) | 94.6 (11.7) | 97.1 (7.36) | 97.3 (5.92)
  Week 11 Day 1, 0 hr (pre-dose) (n=41,10,33,10): number analyzed (Participants) | 41 | 10 | 33 | 10
  Week 11 Day 1, 0 hr (pre-dose) (n=41,10,33,10) | 92.7 (17.8) | 82.3 (30.9) | 97.5 (6.08) | 98.3 (2.39)
  Week 15 Day 1, 0 hr (pre-dose) (n=39,9,33,11): number analyzed (Participants) | 39 | 9 | 33 | 11
  Week 15 Day 1, 0 hr (pre-dose) (n=39,9,33,11) | 92.6 (18.9) | 98.9 (2.90) | 96.8 (8.46) | 92.5 (19.0)
  Week 19 Day 1, 0 hr (pre-dose) (n=36,9,35,10): number analyzed (Participants) | 36 | 9 | 35 | 10
  Week 19 Day 1, 0 hr (pre-dose) (n=36,9,35,10) | 92.4 (12.3) | 83.5 (34.8) | 96.8 (7.36) | 96.7 (5.51)
  Week 23 Day 1, 0 hr (pre-dose) (n=42,11,34,9): number analyzed (Participants) | 42 | 11 | 34 | 9
  Week 23 Day 1, 0 hr (pre-dose) (n=42,11,34,9) | 86.5 (26.3) | 92.0 (13.5) | 94.2 (17.6) | 92.2 (15.7)
  Week 27 Day 1, 0 hr (pre-dose) (n=37,10,33,9): number analyzed (Participants) | 37 | 10 | 33 | 9
  Week 27 Day 1, 0 hr (pre-dose) (n=37,10,33,9) | 87.6 (26.1) | 91.6 (19.4) | 95.4 (10.4) | 87.0 (18.5)
  Week 31 Day 1, 0 hr (pre-dose) (n=36,10,32,9): number analyzed (Participants) | 36 | 10 | 32 | 9
  Week 31 Day 1, 0 hr (pre-dose) (n=36,10,32,9) | 90.9 (18.7) | 89.1 (19.8) | 97.3 (7.02) | 75.5 (37.9)
  Week 35 Day 1, 0 hr (pre-dose) (n=32,11,29,10): number analyzed (Participants) | 32 | 11 | 29 | 10
  Week 35 Day 1, 0 hr (pre-dose) (n=32,11,29,10) | 93.1 (18.0) | 92.8 (10.3) | 92.7 (16.4) | 70.6 (41.0)
  Week 39 Day 1, 0 hr (pre-dose) (n=33,8,33,11): number analyzed (Participants) | 33 | 8 | 33 | 11
  Week 39 Day 1, 0 hr (pre-dose) (n=33,8,33,11) | 85.4 (23.6) | 89.7 (23.6) | 92.7 (18.7) | 89.8 (17.9)
  Week 43 Day 1, 0 hr (pre-dose) (n=31,3,32,8): number analyzed (Participants) | 31 | 3 | 32 | 8
  Week 43 Day 1, 0 hr (pre-dose) (n=31,3,32,8) | 93.1 (15.4) | 99.0 (1.67) | 95.3 (11.0) | 99.1 (2.08)
  Week 47 Day 1, 0 hr (pre-dose) (n=28,2,32,9): number analyzed (Participants) | 28 | 2 | 32 | 9
  Week 47 Day 1, 0 hr (pre-dose) (n=28,2,32,9) | 91.7 (17.7) | 98.8 (1.77) | 95.8 (7.45) | 73.1 (42.4)
  Week 51 Day 1, 0 hr (pre-dose) (n=27,3,26,9): number analyzed (Participants) | 27 | 3 | 26 | 9
  Week 51 Day 1, 0 hr (pre-dose) (n=27,3,26,9) | 86.4 (25.8) | 95.4 (4.24) | 92.5 (19.3) | 93.8 (11.8)

27. Secondary Outcome: Adverse Events by Preferred Term Related to Study Treatment
Description: as for outcome 6
Time Frame: as for outcome 6
Population: Safety analysis set - all treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Age 12 to <18 Years, 5 mg/kg | Age 6 to <12 Years, 5 mg/kg | Age 6 to <12 Years, 8.5 mg/kg | Age 2 to <6 Years, 8.5 mg/kg
Number analyzed (Participants) | 50 | 13 | 40 | 14
Participants
  Number of participants with at least one event | 16 | 5 | 14 | 4
  Infusion related reaction | 5 | 2 | 3 | 1
  Back pain | 3 | 0 | 4 | 2
  Nausea | 3 | 0 | 1 | 0
  Pain in extremity | 2 | 0 | 2 | 0
  Sickle cell anaemia with crisis | 0 | 0 | 2 | 1
  Arthralgia | 0 | 1 | 1 | 0
  Conjunctivitis | 1 | 1 | 0 | 0
  Dizziness | 2 | 0 | 0 | 0
  Headache | 1 | 0 | 1 | 0
  Infusion site pain | 1 | 0 | 1 | 0
  Myalgia | 1 | 1 | 0 | 0
  Neutropenia | 0 | 0 | 1 | 1
  Pain | 1 | 1 | 0 | 0
  Vomiting | 2 | 0 | 0 | 0
  Abdominal pain | 0 | 1 | 0 | 0
  Agitation | 1 | 0 | 0 | 0
  Alopecia | 0 | 0 | 1 | 0
  Anaemia | 0 | 0 | 1 | 0
  Asthenia | 0 | 0 | 1 | 0
  Blood bilirubin increased | 1 | 0 | 0 | 0
  Blood creatine phosphokinase increased | 1 | 0 | 0 | 0
  Dyspnoea | 0 | 1 | 0 | 0
  Fatigue | 1 | 0 | 0 | 0
  Hot flush | 1 | 0 | 0 | 0
  Hypersensitivity | 0 | 0 | 1 | 0
  Malaise | 0 | 1 | 0 | 0
  Muscle fatigue | 1 | 0 | 0 | 0
  Neck pain | 1 | 0 | 0 | 0
  Paraesthesia | 0 | 0 | 1 | 0
  Pruritus | 0 | 1 | 0 | 0
  Pyrexia | 0 | 1 | 0 | 0
  Sacral pain | 0 | 0 | 1 | 0
  Spinal pain | 0 | 0 | 1 | 0
  Vascular access complication | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events are reported from the first dose of study treatment until end of study treatment Week 103 plus 105 days post-treatment follow-up, up to a maximum timeframe of approximately 2 years and 3.25 months.
Groups:
- Age 12 to < 18 Years, 5 mg/kg: Age 12 to < 18 years, 5 mg/kg
- Age 6 to < 12 Years, 5 mg/kg: Age 6 to < 12 years, 5 mg/kg
- Age 6 to < 12 Years, 8.5 mg/kg: Age 6 to < 12 years, 8.5 mg/kg
- Age 2 to < 6 Years, 8.5 mg/kg: Age 2 to < 6 years, 8.5 mg/kg
- All Participants: All Participants / All arms combined / Total
Arm/Group | Age 12 to < 18 Years, 5 mg/kg | Age 6 to < 12 Years, 5 mg/kg | Age 6 to < 12 Years, 8.5 mg/kg | Age 2 to < 6 Years, 8.5 mg/kg | All Participants
All-Cause Mortality (participants affected / at risk) | 1/50 | 0/13 | 0/40 | 0/14 | 1/117
Serious Adverse Events (participants affected / at risk) | 18/50 | 9/13 | 20/40 | 12/14 | 59/117
Other Adverse Events (participants affected / at risk) | 46/50 | 13/13 | 36/40 | 13/14 | 108/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Age 12 to < 18 Years, 5 mg/kg (N=50) | Age 6 to < 12 Years, 5 mg/kg (N=13) | Age 6 to < 12 Years, 8.5 mg/kg (N=40) | Age 2 to < 6 Years, 8.5 mg/kg (N=14) | All Participants (N=117)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 5 | 1 | 9
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
Mesenteric lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Hyperthermia (General disorders) | 0 | 0 | 0 | 1 | 1
Pain (General disorders) | 1 | 0 | 2 | 3 | 6
Pyrexia (General disorders) | 2 | 2 | 1 | 4 | 9
Cholecystitis (Hepatobiliary disorders) | 0 | 2 | 0 | 0 | 2
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 2 | 0 | 3
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 2
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
COVID-19 (Infections and infestations) | 4 | 0 | 1 | 2 | 7
Cellulitis (Infections and infestations) | 0 | 0 | 3 | 0 | 3
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Encephalitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1 | 2
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Meningitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Metapneumovirus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Parainfluenzae virus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Parvovirus B19 infection (Infections and infestations) | 0 | 1 | 1 | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 4 | 3 | 9
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Pneumonia viral (Infections and infestations) | 0 | 0 | 1 | 1 | 2
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Thrombophlebitis septic (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Viral infection (Infections and infestations) | 0 | 0 | 2 | 1 | 3
Brain herniation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Human rhinovirus test positive (Investigations) | 0 | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3 | 4
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 2
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Status migrainosus (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Superficial vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Age 12 to < 18 Years, 5 mg/kg (N=50) | Age 6 to < 12 Years, 5 mg/kg (N=13) | Age 6 to < 12 Years, 8.5 mg/kg (N=40) | Age 2 to < 6 Years, 8.5 mg/kg (N=14) | All Participants (N=117)
Anaemia (Blood and lymphatic system disorders) | 8 | 1 | 4 | 3 | 16
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 2
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 3 | 2 | 6
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 0 | 4
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 4 | 2 | 6
Bundle branch block right (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Right ventricular enlargement (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 1 | 0 | 2
Xerophthalmia (Eye disorders) | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 10 | 5 | 12 | 1 | 28
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 3 | 0 | 4
Constipation (Gastrointestinal disorders) | 9 | 3 | 6 | 2 | 20
Diarrhoea (Gastrointestinal disorders) | 5 | 1 | 5 | 2 | 13
Gastritis (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 3
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 9 | 0 | 5 | 0 | 14
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 14 | 2 | 4 | 1 | 21
Chest pain (General disorders) | 3 | 2 | 4 | 1 | 10
Device related thrombosis (General disorders) | 0 | 1 | 0 | 0 | 1
Fatigue (General disorders) | 3 | 0 | 1 | 0 | 4
Hyperthermia (General disorders) | 0 | 0 | 0 | 1 | 1
Influenza like illness (General disorders) | 2 | 0 | 2 | 1 | 5
Malaise (General disorders) | 0 | 1 | 0 | 0 | 1
Pain (General disorders) | 2 | 3 | 4 | 2 | 11
Pyrexia (General disorders) | 12 | 5 | 16 | 5 | 38
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 3 | 0 | 5
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 0 | 2
COVID-19 (Infections and infestations) | 11 | 1 | 4 | 2 | 18
Conjunctivitis (Infections and infestations) | 1 | 1 | 0 | 1 | 3
Eye infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 3 | 0 | 3 | 0 | 6
Influenza (Infections and infestations) | 2 | 2 | 8 | 0 | 12
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 3 | 5
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 1 | 2
Otitis media (Infections and infestations) | 1 | 0 | 1 | 1 | 3
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 3 | 0 | 5 | 1 | 9
Respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 2 | 4
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 2 | 1 | 1 | 5
Suspected COVID-19 (Infections and infestations) | 3 | 1 | 0 | 0 | 4
Tonsillitis (Infections and infestations) | 1 | 2 | 2 | 1 | 6
Upper respiratory tract infection (Infections and infestations) | 9 | 1 | 2 | 4 | 16
Urinary tract infection (Infections and infestations) | 6 | 1 | 1 | 3 | 11
Viral infection (Infections and infestations) | 0 | 1 | 1 | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 1 | 3
Eye contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 4 | 2 | 3 | 1 | 10
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 2
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | 3
Nasal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Penis injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1 | 2 | 0 | 5
Amylase increased (Investigations) | 0 | 1 | 0 | 0 | 1
Anti factor Xa activity decreased (Investigations) | 0 | 1 | 0 | 0 | 1
Arterial flow velocity increased (Investigations) | 0 | 0 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 2 | 1 | 0 | 6
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 0 | 1 | 3
Blood bilirubin increased (Investigations) | 3 | 1 | 1 | 0 | 5
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 1 | 2
C-reactive protein increased (Investigations) | 0 | 0 | 1 | 2 | 3
Cardiac murmur (Investigations) | 0 | 1 | 1 | 0 | 2
Epstein-Barr virus test positive (Investigations) | 0 | 1 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0 | 1
Influenza A virus test negative (Investigations) | 0 | 1 | 0 | 0 | 1
Influenza virus test negative (Investigations) | 0 | 1 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 1 | 1 | 0 | 0 | 2
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 1
Polymerase chain reaction negative (Investigations) | 0 | 1 | 0 | 0 | 1
SARS-CoV-2 test negative (Investigations) | 12 | 3 | 0 | 0 | 15
SARS-CoV-2 test positive (Investigations) | 3 | 0 | 0 | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 3
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 1 | 7 | 1 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 2 | 9 | 4 | 26
Bone infarction (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 3
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 1 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 0 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1 | 4
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 4 | 0 | 3 | 0 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 3 | 10 | 3 | 27
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 2
Dizziness (Nervous system disorders) | 5 | 1 | 1 | 0 | 7
Headache (Nervous system disorders) | 19 | 4 | 10 | 3 | 36
Anxiety (Psychiatric disorders) | 4 | 0 | 1 | 0 | 5
Insomnia (Psychiatric disorders) | 3 | 0 | 0 | 0 | 3
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 3 | 0 | 0 | 0 | 3
Haematuria (Renal and urinary disorders) | 3 | 0 | 0 | 0 | 3
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Asthma exercise induced (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 9 | 5 | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1 | 1 | 8
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2 | 0 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1 | 0 | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 2 | 2 | 10
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1 | 0 | 0 | 5
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0 | 4
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 0 | 0 | 2 | 4
Pallor (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-03-14): https://cdn.clinicaltrials.gov/large-docs/65/NCT03474965/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-15): https://cdn.clinicaltrials.gov/large-docs/65/NCT03474965/SAP_001.pdf